CLINICAL TRIAL: NCT02894177
Title: Is Transcutaneous Carbon Dioxide Pressure (tcPCO2) Monitoring During Spontaneous Breathing Trials Useful to Predict Extubation Failure in Mechanically Ventilated Patients in the ICU?
Brief Title: Transcutaneous Carbon Dioxide Pressure (tcPCO2) Monitoring for the Prediction of Extubation Failure in the ICU
Acronym: tcPCO2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Versailles Hospital (Other)
Responsible Party: Principal Investigator, Henao Juliana, study coordinator, Versailles Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: P15/07_ tcPCO2
Record Dates: First submitted 2016-08-14; First posted 2016-09-09 (Estimated); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Ventilator Weaning
Keywords: E02.880.820.950

STUDY DESIGN:
Intervention Model Description: tcPCO2 will be monitored in all patients performing SBTs. The difference between maximal and initial tcPCO2 (ΔtcPCO2) in patients succeeding extubation will be compared with ΔtcPCO2 in patients failing extubation.
Masking Description: Care providers will be blinded of tcPCO2 measurements to avoid influencing extubation decisions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- tcPCO2 measurement arm (Experimental): Patients will be monitored by tcPCO2 during spontaneous breathing trials
  Interventions: Procedure: tcPCO2 measurement

INTERVENTIONS:
Procedure: tcPCO2 measurement — tcPCO2 continuous monitoring during spontaneous breathing trials

SUMMARY:
Difficult weaning from ventilation and extubation failure are major issues in intensive care, concerning 30% and 12% of patients respectively. These can be partly explained by the lack of accuracy of spontaneous breathing trial (SBT) failure criteria to predict extubation failure. The investigators performed a pilot study to evaluate transcutaneous carbon dioxide pressure (tcPCO2) monitoring during SBTs. The results showed that the difference between maximum and initial tcPCO2 (or ΔtcPCO2) was significantly higher in the group of patients who failed SBTs according to the usual criteria. Moreover, the results suggested that ΔtcPCO2 could be an accurate and early criterion for SBT failure. The size of the study could not examine ΔtcPCO2 regarding extubation failure. Therefore, the main objective of this study is to determine if Δ tcPCO2 during SBTs is associated with extubation failure.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years old,
* ICU indicated
* invasive mechanical ventilation via orotracheal or nasotracheal intubation
* presence of criteria for initiation of the weaning process as stated on our ICU's protocol
* resolution of the disease leading to mechanical ventilation

Exclusion Criteria:

* mechanical ventilation during less than 24 hours
* Tracheotomy and tracheostomy at ICU admission
* Pregnancy
* Patient under legal protection

  * Patient enrolled in another study regarding weaning or CO2 metabolism

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2017-09-04 (Actual); Primary Completion 2020-04-02 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Difference between maximum and initial tcPCO2 (ΔtcPCO2) during SBTs in patients who fail extubation compared to patients who have been successfully extubated. | 7 days
  Extubation failure: need for reintubation, rescue non invasive ventilation or death within 7 days following extubation

SECONDARY OUTCOMES:
Association between ΔtcPCO2 and extubation failure after adjustment on post extubation ventilation protocols (preventive non invasive ventilation or preventive Optiflow) | 7 days
  Different post-extubation ventilation protocols may include preventive non invasive ventilation or Optiflow.
Association between extubation decisions and ΔtcPCO2. | 1 week
Adverse Events associated with tcPCO2 monitoring. | 1 week
Optimal ΔtcPCO2 threshold to predict extubation failure by a ROC curve. | 7 days
Compare ROC curves obtained by different extubation failure predictors | 7 days
  ROC curves obtained with:
  * usual SBT failure criteria
  * deltatcPCO2 alone
  * usual criteria and ΔtcPCO2 combined
  * shallow breathing index
  * shallow breathing index and ΔtcPCO2 combined
  * ΔtcPCO2, shallow breathing index and usual SBT failure criteria combined
Determine if ΔtcPCO2 is an early predictor of extubation failure (happening before other criteria of failed SBT) | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Henao-Brasseur Juliana, Principal Investigator — CH Versailles
Locations (1):
- CH Versailles, Le Chesnay, France

IPD SHARING:
Plan to Share IPD: No